CLINICAL TRIAL: NCT06327698
Title: Efficacy and Safety of Cadonilimab in Combination With Anlotinib in the Treatment of Locally Progressive or Metastatic Melanoma With First-Line Therapy Failure: A Single-arm, Open-label, Multicenter Phase II Clinical Study
Brief Title: Cadonilimab in Combination With Anlotinib in the Treatment of Locally Progressive or Metastatic Melanoma With First-Line Therapy Failure
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-C-S-0010
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Melanoma
Keywords: locally advanced or metastatic melanoma; cadonilimab; anlotinib; First-Line Therapy Failure
MeSH Terms: conditions — Melanoma | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination+ Anlotinib (Experimental): Cadonilimab (AK104) (10 mg/kg, Q3W, administered on the frst day of each cycle, Q3W, until there is no clinical beneft) + anlotinib (8 mg, QD, 2 weeks off for 1 week)
  Interventions: Drug: Cadonilimab; Drug: anlotinib

INTERVENTIONS:
Drug: Cadonilimab — Injectable solution
  Other Names: AK104
Drug: anlotinib — capsule

SUMMARY:
This study is an open-label, multicenter, single-arm Phase II clinical study to evaluate the effectiveness of cadonilimab (AK104) in combination with anlotinib in the treatment of locally advanced or metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years and ≤ 75 years
2. Has a histologically confrmed diagnosis of malignant melanoma
3. Previously received failed first-line treatment for melanoma
4. Patients may have a history of liver metastases, but the metastases should be less than 3
5. Patients with treatment-asymptomatic brain metastases may be included, must be free of disease progression on computed tomography (CT) or magnetic resonance imaging (MRI), stable for at least 3 months, and free of steroid medication for at least 4 weeks
6. Those with at least 1 measurable lesion (RECIST version 1.1)
7. ECOG 0-1
8. Non-lactating patients
9. Good organ function

Exclusion Criteria:

1. Previous (within 5 years) or concurrent other malignant tumors, except for cured local tumors (such as basal cell skin cancer, squamous cell skin cancer, superficial bladder cancer, cervical carcinoma in situ, breast carcinoma in situ, etc.) and breast cancer without recurrence > 3 years after radical resection
2. Has an active or potentially recurrent autoimmune disease
3. History of severe allergic reaction to any monoclonal antibody and/or component of the study drug
4. Known presence of active tuberculosis TB
5. Currently receiving cancer treatment (chemotherapy, radiotherapy, immunotherapy, or biologic therapy)
6. Received a live vaccine within 30 days prior to the first dose, or plans to receive a live vaccine during the study
7. Known history of psychiatric illness, substance abuse, alcoholism, or drug abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Response Rate | from the frst drug administration up to two years
  ORR is the proportion of patients with best response of complete response (CR) and PR

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | from the frst drug administration up to two years
  Time from the date of frst study treatment administration to the date of first
Disease Control Rate (DCR) | from the frst drug administration up to two years
  Proportion of patients whose best overall response is either CR, PR, or SD
Safety and tolerability | from the frst drug administration up to two years
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE